CLINICAL TRIAL: NCT04359030
Title: In Vivo Calcium Score Measurement After Freestyle Full Root Replacement in Young Adults
Brief Title: Freestyle-Perimount Calcification Comparison
Status: Completed | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Matteo Pettinari, Principal Investigator, Ziekenhuis Oost-Limburg
Other Study IDs: ctu2020003
Record Dates: First submitted 2020-03-17; First posted 2020-04-24 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Aortic Valve Disease; Valve Heart Disease
MeSH Terms: conditions — Aortic Valve Disease; Heart Valve Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Freestyle group: Patients treated with a Freestyle aortic valve bioprosthesis
  Interventions: Diagnostic Test: Multislice CT scanning for aortic wall calcification; Diagnostic Test: Transthoracic stress echocardiography
- Perimount group: Patients treated with a Perimount aortic valve bioprosthesis
  Interventions: Diagnostic Test: Multislice CT scanning for aortic wall calcification; Diagnostic Test: Transthoracic stress echocardiography

INTERVENTIONS:
Diagnostic Test: Multislice CT scanning for aortic wall calcification — Multislice CT scanning for aortic wall calcification
Diagnostic Test: Transthoracic stress echocardiography — Transthoracic stress echocardiography

SUMMARY:
The aim of this study is to evaluate the rate and anatomy of the aortic wall and leaflet calcification of the FS prosthesis implanted as full root in patients younger than 60 years compared to a stented bioprostheses (Perimount Magna Ease, PM). A 3D CT scan will be used to assess the calcification score and to determine the relationship between calcification and aortic valve leaflet.

DETAILED DESCRIPTION:
A recent update of the American Hear Association and American College of Cardiology Guidelines for the Management of Patients With Valvular Heart Disease1 recommended that for patients between 50 and 70 years of age, it is reasonable to the choice of either a mechanical or bioprosthetic valve; the threshold for biological valves continues to decrease and more younger adults will receive this kind of prosthesis. However the best biological option for these patients is still a matter of debate. Stented bio-prosthesis is the most common choice. However, the predicted 15-year risk of needing reoperation because of structural deterioration is 22% for patients 50 years of age2.

In the late 80's stentless valve as the Medtronic Freestyle (FS) has been introduced with the hope that it may provide physiological flow in the aortic root, sinuses, and coronary orifices and a low risk of thromboembolism. Several randomized study and meta-analysis demonstrated improved hemodynamic, a larger orifice area and a midterm survival advantage of stentless aortic valve compared to stented aortic valve replacement3, 4. The FS valve is believed to provide greater durability and superior hemodynamic performance due to the low mechanical stress on the leaflet tissues. The failure mode of the FS is thought to be mostly calcification of the aorta wall and cusp tears because collagen degradation5. This phenomenon is inflammation mediated process.

Aim of this study is to evaluate the rate and anatomy of the aortic wall and leaflet calcification of the FS prosthesis implanted as full root in patients younger than 60 years compared to a stented bioprostheses (Perimount Magna Ease, PM). A 3D CT scan will be used to assess the calcification score and to determine the relationship between calcification and aortic valve leaflet.

Between 2007 and 2017, among patients younger than 60 years of age, 51 patients underwent a full root replacement with a FS and 49 received a Perimount Magna Ease prosthesis. Those patients will undergo a 3D CT scan. The group of the patient with PM will be matched in function of age and interval of follow-up with the FS group.

A transthoracic echocardiogram will be performed to check residual valve insufficiency and trans-valvular gradients. A cardiopulmonary exercise test ( with extraction of maximal oxygen consumption ) combined with a trans thoracic echocardiography (stress echocardiography) will be performed to evaluate the patients exercise capacity and its influence on the cardiac and valve function.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Patients treated with FS or PM
* Age less than 60 at the moment of the implant

Exclusion Criteria:

* Kidney failure or contrast allergy
* Previous endocarditis and aortic dissection
* Pregnancy or lactation

Max Age: 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Patients operated for aortic valve stenosis at least three years earlier undergoing a valve replacement with Freestyle (FS) or Perimount (PM) bioprosthesis under the age of 60 years.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Quantification of aortic leaflet Calcium-score in FS and PM valve | 3 years
  The Agatston score. The score is calculated using a weighted value assigned to the highest density of calcification in a given coronary artery. The density is measured in Hounsfield units (HU), and score of 1 for 130-199 HU, 2 for 200-299 HU, 3 for 300-399 HU, and 4 for 400 HU and greater. The higher the score the more the calcification.

SECONDARY OUTCOMES:
Echocardiographic function of the aortic valve at rest and during exercise: transvalvular mean and peak gradient | 3 years
  Aortic valve mean and peak gradient: mmHg
Echocardiographic function of the aortic valve at rest and during exercise: Valve regurgitation | 3 years
  Aortic valve regurgitation: vena contracta (mm)
Exercise capacity: New York Heart Association class | 3 years
  New York Heart Association class from 1 to 4 with 1=no dyspnea during exercise till 4= dyspnea in rest;
Exercise capacity: maximum oxygen consumption | 3 years
  max oxygen consumption measured in ml/kg*min

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Pettinari, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost Limburg, Genk, Limburg, Belgium